CLINICAL TRIAL: NCT00636818
Title: An Open Study of Atomoxetine (LY139603) in Adult Subjects With Attention-deficit/Hyperactivity Disorder
Brief Title: Atomoxetine Asian Study in Adult Subjects With Attention-Deficit/Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12112; B4Z-JE-LYEH (Other: Eli Lilly and Company)
Record Dates: First submitted 2008-03-07; First posted 2008-03-14 (Estimated); Results first posted 2009-12-23 (Estimated); Last update posted 2010-11-04 (Estimated); Status verified 2010-10

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Atomoxetine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Atomoxetine (Experimental)
  Interventions: Drug: Atomoxetine

INTERVENTIONS:
Drug: Atomoxetine — Study drug is administered once daily in the morning. This study is designed with 4-step titration. At Day 1, study drug is started from 40 mg/day, and is increased to 80 mg/day on Day 7, 105 mg/day on Day 14, and 120 mg/day on Day 28. Total administration period is 8 weeks. The dosage is adjusted according to investigator's decision based on safety and tolerability.
  Other Names: LY139603; Strattera

SUMMARY:
The primary objective of this clinical study is to assess overall safety and tolerability as measured by discontinuation rate due to adverse events in doses up to 120 mg/day in relation to global clinical studies in adult subjects who meet Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV™) criteria for Attention-Deficit/Hyperactivity Disorder (ADHD).

ELIGIBILITY:
Inclusion Criteria:

1. at least 18 years of age
2. meet Conners' Adult ADHD Diagnostic Interview for DSM-IV (CAADID) diagnostic criteria for current ADHD as well as meeting criteria for a historical diagnosis of ADHD during childhood
3. have a Clinical Global Impressions-ADHD-Severity (CGI-ADHD-S) score of 4 (moderate symptoms) or greater

Exclusion Criteria:

1. Patients who meet DSM-IV diagnostic criteria for current major depression and also patients who have total score of more than 12 on the 17-item Hamilton Depression Rating Scale (HAMD-17) at Visit 1 and Visit 2. Patients who have both a current or past history of major depression and have received any anti-depression drug therapy within 6 months of Visit 1.
2. Patients who meet DSM-IV diagnostic criteria for have a current anxiety disorder and also require anti-anxiety drug therapy except for those taking benzodiazepines analogues for anxiety which need to be limited.
3. Patients who have any history of bipolar disorder (DSM-IV) , any history of schizophrenia or any history of a psychotic disorder (DSM-IV) will be excluded from the study.
4. Patients who have been diagnosed (DSM-IV) with a pervasive developmental disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2008-03; Primary Completion 2008-09 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) Mon - Fri 9 AM - 5PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (11):
- China (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Beijing
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Changsha
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Guangzhou
- South Korea (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Busan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Incheon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jeonju
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seoul
- Taiwan (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Neihu Taipei
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Niao Sung Hsiang
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taipei
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taoyuan District

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Atomoxetine
Started | 45
Received at Least One Dose of Study Drug | 44 (One patient was lost to follow up and did not receive any study drug.)
Completed | 34
Not Completed | 11
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 2
Not completed — Entry Criteria Exclusion | 3
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Arm/Group | Atomoxetine
Number analyzed (Participants) | 44
Age Continuous [Mean (Standard Deviation); unit: years] | 28.24 (9.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 30
Region of Enrollment [Number; unit: participants]
  Taiwan | 12
  China | 15
  Korea, Republic of | 17
Attention-Deficit/Hyperactivity Disorder (ADHD) Subtype [Number; unit: participants]
  Inattentive | 25
  Hyperactive/Impulsive | 2
  Mixed | 17
Prior Stimulant Exposure [Number; unit: participants]
  No | 30
  Yes | 13
  Unknown | 1
Race/Ethnicity [Number; unit: participants]
  East Asian | 44
Height [Mean (Standard Deviation); unit: centimeters (cm)] | 168.98 (6.04)
Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 64.53 (9.27)

OUTCOME MEASURES:

1. Primary Outcome: Discontinuations Due to Adverse Events (AE)
Description: The definition of a study adverse event was any unfavorable medical event, newly emerged or a deterioration of a preexisting condition, in other words any untoward medical occurrence in a patient administered a pharmaceutical product, without regard to the possibility of a causal relationship, that occurred after the visit for informed consent and up to the visit for completion of administration, or discontinuation.
Time Frame: Baseline to 8 Weeks
Population: Number of participants who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Atomoxetine
Number analyzed (Participants) | 44
participants
  Participants with >=1 AE (Discontinuation) | 1
  Somnolence (Nervous System Disorder) | 1

2. Secondary Outcome: Change From Baseline to 8 Week Endpoint in Conners' Adult Attention-Deficit/Hyperactivity Disorder (ADHD) Rating Scale-Investigator Rated:Screening Version (CAARS-Inv:SV) Total ADHD Symptom Score
Description: Conners' Adult Attention-Deficit Hyperactivity Disorder (ADHD) Rating Scale-Investigator Rating:Screening Version. Total ADHD symptom score consisted of 18 items (sum of inattention and hyperactivity-impulsivity subscales) using a 4-point scale (0=not at all/never to 3=very much/very frequently) for total score range of 0 to 54.
Time Frame: Baseline and 8 Weeks
Population: Number of participants who received at least one dose of study drug and had a baseline and at least one post-baseline value. Last observation carried forward.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomoxetine
Number analyzed (Participants) | 43
units on a scale
  Baseline | 32.0 (6.3)
  Change from Baseline | -12.8 (10.4)
Statistical Analysis 1: Comparison: Atomoxetine; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — P-value for Change from Baseline. Change=Endpoint minus Baseline

3. Secondary Outcome: Change From Baseline to 8 Week Endpoint in Clinical Global Impressions-ADHD Severity (CGI-ADHD-S)
Description: Measures severity of the patient's overall severity of ADHD symptoms (1=normal, not at all ill; 7=among the most extremely ill patients).
Time Frame: Baseline and 8 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomoxetine
Number analyzed (Participants) | 43
units on a scale
  Baseline | 4.8 (0.8)
  Change from Baseline | -1.7 (1.3)
Statistical Analysis 1: Comparison: Atomoxetine; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — P-value for Change from Baseline. Change=Endpoint minus Baseline

4. Secondary Outcome: Change From Baseline to 8 Week Endpoint in Conners' Adult ADHD Rating Scale-Self Rated:Screening Version (CAARS-S:SV) Total ADHD Symptom Score
Description: Conners' Adult Attention-Deficit Hyperactivity Disorder (ADHD) Rating Scale-Self Rating:Screening Version. Total ADHD symptom score consisted of 18 items (sum of inattention and hyperactivity-impulsivity subscales) using a 4-point scale (0=not at all/never to 3=very much/very frequently) for total score range of 0 to 54.
Time Frame: Baseline and 8 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomoxetine
Number analyzed (Participants) | 43
units on a scale
  Baseline | 30.6 (9.7)
  Change from Baseline | -12.1 (10.2)
Statistical Analysis 1: Comparison: Atomoxetine; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — P-value for Change from Baseline. Change=Endpoint minus Baseline

5. Secondary Outcome: Change From Baseline to 8 Week Endpoint in 17-Item Hamilton Depression Rating Scale (HAMD-17)
Description: The 17-item HAMD measures depression severity. Each item was evaluated and scored using either a 5-point scale (e.g. absent, mild, moderate, severe, very severe) or a 3-point scale (e.g. absent, mild, marked). The total score of HAMD-17 may range from 0 (normal) to 52 (severe).
Time Frame: Baseline and 8 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomoxetine
Number analyzed (Participants) | 42
units on a scale
  Baseline | 4.8 (3.9)
  Change from Baseline | -1.5 (3.8)
Statistical Analysis 1: Comparison: Atomoxetine; Test type: Superiority or Other; p = 0.013, t-test, 2 sided — P-value for Change from Baseline. Change=Endpoint minus Baseline

6. Secondary Outcome: Change From Baseline to 8 Week Endpoint in Hamilton Anxiety Rating Scale (HAMA-14)
Description: The HAMA-14 scale measures anxiety symptoms accompanying Major Depressive Disorder (MDD). Each item of the 14-item HAMA was scored from 0 (not present) to 4 (very severe), with a resulting maximum total score of 56.
Time Frame: Baseline and 8 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomoxetine
Number analyzed (Participants) | 42
units on a scale
  Baseline | 6.7 (4.7)
  Change from Baseline | -2.0 (4.4)
Statistical Analysis 1: Comparison: Atomoxetine; Test type: Superiority or Other; p = 0.005, t-test, 2 sided — P-value for Change from Baseline. Change=Endpoint minus Baseline

7. Secondary Outcome: Change From Baseline to 8 Week Endpoint in Stroop Color Word Test
Description: This was a psychological test to observe the interference in which disparity between the meaning and color affects reading speed. A subject was given 3 tasks of recognition: reading the printed colored ink (Color Test), reading color words in black ink (Word Test), and interference, reading color words printed in different colored ink (Word-Color Test). The test was scored on the number of correct answers. There were 100 items for each of the three categories and if they made it through the 100 words with time remaining, they would repeat the list.
Time Frame: Baseline and 8 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: number of correct answers
Arm/Group | Atomoxetine
Number analyzed (Participants) | 42
number of correct answers
  Word Test: Baseline | 82.4 (16.6)
  Word Test: Change from Baseline | 4.5 (9.9)
  Color Test: Baseline | 68.7 (14.8)
  Color Test: Change from Baseline | 4.8 (10.6)
  Color-Word Test: Baseline | 49.0 (16.5)
  Color-Word Test: Change from Baseline | 3.5 (15.4)
Statistical Analysis 1: Comparison: Atomoxetine; Test type: Superiority or Other; p = 0.005, t-test, 2 sided — P-value for Word Test: Change from Baseline. Change=Endpoint minus Baseline
Statistical Analysis 2: Comparison: Atomoxetine; Test type: Superiority or Other; p = 0.005, t-test, 2 sided — P-value for Color Test: Change from Baseline. Change=Endpoint minus Baseline
Statistical Analysis 3: Comparison: Atomoxetine; Test type: Superiority or Other; p = 0.144, t-test, 2 sided — P-value for Color-Word Test: Change from Baseline. Change=Endpoint minus Baseline

8. Secondary Outcome: Change From Baseline to 8 Week Endpoint in Short Form-36 Version 2 (SF-36v2)
Description: SF-36 assesses quality of life (QoL) on 8 domains and 2 summary scores (mental component summary [MCS] and physical component summary [PCS]). MCS and PCS scores=0-100 (higher scores indicate better QoL). Raw domain scores: general health=5-25; physical functioning=10-30; role-physical=4-20; role-emotional=3-15; social functioning=2-10; bodily pain=2-12; vitality=4-20; mental health=5-25. Using norm based scores, all domains, MCS and PCS scores have average score of 50 with standard deviation of 10. Norm-based score=Z-score*10+50 in each subscale. Range cannot be specified in norm-based scores.
Time Frame: Baseline and 8 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: T-Score
Arm/Group | Atomoxetine
Number analyzed (Participants) | 42
T-Score
  Physical Component Summary: Baseline | 46.77 (9.11)
  Physical Component Summary: Change from Baseline | -0.38 (9.23)
  Mental Component Summary: Baseline | 43.71 (6.93)
  Mental Component Summary: Change from Baseline | 3.62 (5.36)
  Physical Functioning: Baseline | 53.12 (6.79)
  Physical Functioning: Change from Baseline | -3.02 (9.09)
  Role-Physical: Baseline | 43.58 (11.36)
  Role-Physical: Change from Baseline | 1.30 (10.94)
  Bodily Pain: Baseline | 50.46 (10.71)
  Bodily Pain: Change from Baseline | 1.32 (9.31)
  General Health Perception: Baseline | 47.81 (9.67)
  General Health Perception: Change from Baseline | 2.48 (9.17)
  Vitality: Baseline | 43.73 (8.63)
  Vitality: Change from Baseline | 2.78 (8.61)
  Social Functioning: Baseline | 40.97 (11.36)
  Social Functioning: Change from Baseline | 2.82 (10.39)
  Role-Emotional: Baseline | 36.63 (11.59)
  Role-Emotional: Change from Baseline | 5.46 (13.05)
  Mental Health: Baseline | 40.38 (9.42)
  Mental Health: Change from Baseline | 5.51 (8.04)
Statistical Analysis 1: Comparison: Atomoxetine; Test type: Superiority or Other; p = 0.791, t-test, 2 sided — P-value for Physical Component Summary: Change from Baseline. Change=Endpoint minus Baseline
Statistical Analysis 2: Comparison: Atomoxetine; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — P-value for Mental Component Summary: Change from Baseline. Change=Endpoint minus Baseline
Statistical Analysis 3: Comparison: Atomoxetine; Test type: Superiority or Other; p = 0.037, t-test, 2 sided — P-value for Physical Functioning: Change from Baseline. Change=Endpoint minus Baseline
Statistical Analysis 4: Comparison: Atomoxetine; Test type: Superiority or Other; p = 0.446, t-test, 2 sided — P-value for Role-Physical: Change from Baseline. Change=Endpoint minus Baseline
Statistical Analysis 5: Comparison: Atomoxetine; Test type: Superiority or Other; p = 0.365, t-test, 2 sided — P-value for Bodily Pain: Change from Baseline. Change=Endpoint minus Baseline
Statistical Analysis 6: Comparison: Atomoxetine; Test type: Superiority or Other; p = 0.087, t-test, 2 sided — P-value for General Health Perception: Change from Baseline. Change=Endpoint minus Baseline
Statistical Analysis 7: Comparison: Atomoxetine; Test type: Superiority or Other; p = 0.043, t-test, 2 sided — P-value for Vitality: Change from Baseline. Change=Endpoint minus Baseline
Statistical Analysis 8: Comparison: Atomoxetine; Test type: Superiority or Other; p = 0.086, t-test, 2 sided — P-value for Social Functioning: Change from Baseline. Change=Endpoint minus Baseline
Statistical Analysis 9: Comparison: Atomoxetine; Test type: Superiority or Other; p = 0.010, t-test, 2 sided — P-value for Role-Emotional: Change from Baseline. Change=Endpoint minus Baseline
Statistical Analysis 10: Comparison: Atomoxetine; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — P-value for Mental Health: Change from Baseline. Change=Endpoint minus Baseline

9. Secondary Outcome: Number of Participants With Potentially Clinically Significant Changes in Vital Signs During the Study
Description: Vital signs reported are Pulse (beats per minute [bpm]), Systolic Blood Pressure (SBP) (mmHg), and Diastolic Blood Pressure (DBP) (mmHg).
Time Frame: Baseline to 8 Weeks
Population: Number of participants with baseline and post-baseline values.
Measure: Number; unit: participants
Arm/Group | Atomoxetine
Number analyzed (Participants) | 44
participants
  High Pulse (bpm)=Increase ≥15 to a value >120 | 0
  Low Pulse (bpm)=Decrease ≥15 to a value <50 | 0
  High SBP (mmHg)=Increase ≥20 to a value >180 | 0
  Low SBP (mmHg)=Decrease ≥20 to value of at most 90 | 1
  High DBP (mmHg)=Increase ≥15 to value at least 105 | 0
  Low DBP (mmHg)=Decrease ≥15 to value of at most 50 | 0

10. Secondary Outcome: Significant Changes in Body Weight During the Study
Description: Potentially clinically significant weight loss was defined as any decrease of at least 7 percent (%). Potentially clinically significant weight gain was defined as any increase of at least 7%.
Time Frame: Baseline to 8 Weeks
Population: Number of participants with baseline and post-baseline values.
Measure: Number; unit: participants
Arm/Group | Atomoxetine
Number analyzed (Participants) | 44
participants
  Weight Loss = Any Decrease of at Least 7% | 5
  Weight Gain = Any Increase of at Least 7% | 0

11. Secondary Outcome: Number of Participants With Abnormal QTc Interval Based on International Conference on Harmonisation Criterion
Description: The Fridericia correction of the QT interval (QTcF) was used.
Time Frame: Baseline to 8 Weeks
Population: Number of participants with baseline and post-baseline values.
Measure: Number; unit: participants
Arm/Group | Atomoxetine
Number analyzed (Participants) | 42
participants
  QTcF Interval of >450 milliseconds (msec) | 0
  QTcF Interval of >480 msec | 0
  QTcF Interval of >500 msec | 0
  QTcF Interval Increase from Baseline of ≥30 msec | 1
  QTcF Interval Increase from Baseline of ≥60 msec | 0

12. Secondary Outcome: Cytochrome P450 2D6 (CYP2D6) Phenotype Status
Description: CYP2D6 is the primary atomoxetine metabolizing enzyme. Metabolizzer status was determined by focusing on the normal, decreased, and defective allele. Poor metabolizer = defective/defective. Extensive metabolizer is all except for poor metabolizer.
Time Frame: 8 Weeks
Population: Number of participants who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Atomoxetine
Number analyzed (Participants) | 44
participants
  Extensive Metabolizer | 44
  Poor Metabolizer | 0

ADVERSE EVENTS:
Arm/Group | Atomoxetine
Serious Adverse Events (participants affected / at risk) | 1/44
Other Adverse Events (participants affected / at risk) | 41/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atomoxetine (N=44)
Hand-foot-and-mouth disease (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atomoxetine (N=44)
Palpitations (Cardiac disorders) | 5 (6)
Dry mouth (Gastrointestinal disorders) | 5 (5)
Nausea (Gastrointestinal disorders) | 16 (19)
Vomiting (Gastrointestinal disorders) | 4 (5)
Asthenia (General disorders) | 4 (4)
Fatigue (General disorders) | 6 (6)
Irritability (General disorders) | 3 (3)
Anorexia (Metabolism and nutrition disorders) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 7 (8)
Dizziness (Nervous system disorders) | 15 (19)
Headache (Nervous system disorders) | 5 (5)
Somnolence (Nervous system disorders) | 13 (13)
Insomnia (Psychiatric disorders) | 7 (7)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days